CLINICAL TRIAL: NCT05885750
Title: The Impact of Plant-Based Protein-rich Food Products With Varying Degree of Processing on the Human Gut Microbiome Composition and Human Metabolome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Marko Kalliomäki, MD, Clinical Professor, University of Turku
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Newplant
Record Dates: First submitted 2023-05-17; First posted 2023-06-02 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Metabolism; Gut Microbiota; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Airway Resistance

STUDY DESIGN:
Intervention Model Description: Crossover trial with two one-week wash-out periods in-between three interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet 1 (Experimental): Unprocessed or minimally processed plant-based protein-rich food products
  Interventions: Behavioral: Unprocessed
- Diet 2 (Experimental): Mildly processed plant-based protein-rich food products
  Interventions: Behavioral: Mildly processed
- Diet 3 (Experimental): Heavily refined plant-based protein-rich food products
  Interventions: Behavioral: Heavily refined

INTERVENTIONS:
Behavioral: Unprocessed — Participants will consume unprocessed or minimally processed commercially available plant-based protein-rich foods as meat replacement in their normal diet for one week.
  Arms: Diet 1
Behavioral: Mildly processed — Participants will consume mildly processed commercially available plant-based protein-rich foods as meat replacement in their normal diet for one week.
  Arms: Diet 2
Behavioral: Heavily refined — Participants will consume heavily refined processed commercially available plant-based protein-rich foods as meat replacement in their normal diet for one week.
  Arms: Diet 3

SUMMARY:
It is observed that replacing meat with protein-rich plant-based food products are associated with lower mortality and obesity prevention. Sources of plant proteins typically undergo several processing and refinement procedures to improve the taste and digestibility of plant-based food products. These procedures alter the chemical composition, which can impact the nutritional quality of the processed food. It is not known what is the impact of processed products on human metabolism and intestinal microbiota. Therefore, the impact of a set of plant-based protein-rich food products with varying degree of processing on the composition and function of human gut microbiome and metabolism will be assessed in a clinical intervention

DETAILED DESCRIPTION:
Plant-based diets are known to have beneficial effects on both the environment and human health. Replacing animal protein with plant protein reduces overall mortality risk, and replacing meat with legumes and other sources of plant protein can lower the risk of chronic diseases such as type 2 diabetes and cardiovascular disease. However, the benefits of plant protein products is not evident. In order to make plant protein products more palatable and digestible, plant raw materials may go through several processing and refinement procedures. Typically, during these phases, carbohydrate fractions (e.g. dietary fiber) are removed from the plant material, which results in the loss of micronutrients as well as secondary plant metabolites with potentially health effects (e.g. polyphenolic compounds). Salt and various fats are added to some products, which can reduce the nutritional quality of the product. Subsequently, not all plant-based protein-rich foods are automatically healthy as there may be significant differences in the nutritional quality of the processed products, depending on the food processing utilized. Only little research information is available on the effects of processed plant protein products on human metabolism and intestinal microbiota. Therefore, this cross-over clinical intervention will be conducted with 38 healthy participants to investigate the impact of a set of plant-based protein-rich food products with varying degree of processing on the composition and function of human gut microbiome and metabolism will be assessed in a clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* 18-65-years olf
* BMI 18.5-27 kg/m2

Exclusion Criteria:

* Chronic disease with continuous medication
* Antibiotic use in the past 6 months
* Active smoker
* Gluten-free or vegan diet
* Pregnancy, lactation
* Abnormal thyroid, liver, or kidney function
* Low hemoglobin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | one week between the start and end of each intervention
  The changes in metabolism evoked by the interventions
Transcriptomics | one week between the start and end of each intervention
  The changes in endogenous gene expression on RNA level
Metagenomics | one week between the start and end of each intervention
  The alterations in the composition of gut microbiota
Inflammation status by inflammatory cytokines | one week between the start and end of each intervention
  The changes in inflammatory cytokines
Inflammation status by high-sensitive CRP | one week between the start and end of each intervention
  The changes in high-sensitive CRP by clinical biochemistry analysis

SECONDARY OUTCOMES:
Glucose homeostasis | one week between the start and end of each intervention
  Fasting plasma glucose and insulin concentrations by clinical biochemistry analyses
Lipid homeostasis | one week between the start and end of each intervention
  Cholesterol and triglyceride concentrations by clinical biochemistry analyses
Body weight | five weeks (baseline and at the end of the complete study / after three interventions and 2 wash-outs)
  Body weight in kilograms measured by standard weight scale

CONTACTS AND LOCATIONS:
Overall Officials: Kati Hanhineva, PhD, Principal Investigator — University of Turku
Locations (1):
- Food Sciences Unit, Department of Life Technologies, Faculty of Technology, University of Turku, Turku, Finland